CLINICAL TRIAL: NCT06197282
Title: Impact of COVID-19 on Surgical Outcomes in Acute Care Service in a Community Hospital
Brief Title: Impact of COVID-19 on Surgical Outcomes
Status: Completed | Type: Observational
Sponsor: Kern Medical Center (Other)
Responsible Party: Principal Investigator, Amber Jones, Principal Investigator, DO, MPH, Kern Medical Center
Other Study IDs: 22152
Record Dates: First submitted 2024-01-05; First posted 2024-01-09 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: COVID-19; Surgical Outcomes; Postoperative Complications
Keywords: Postoperative outcomes; COVID-19
MeSH Terms: conditions — COVID-19; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 Positive, Symptomatic: Patients undergoing major surgery with a documented positive COVID19 test with in 1 year of surgery and were symptomatic for COVID19 at the time of testing.
  Interventions: Procedure: Major surgery involving general anesthesia
- COVID-19 Positive, Asymptomatic: Patients undergoing major surgery with a documented positive COVID19 test with in 1 year of surgery and were asymptomatic for COVID19 at the time of testing as well as at the time of surgery.
  Interventions: Procedure: Major surgery involving general anesthesia
- Control: COVID-19 Negative: Patients undergoing major surgery with documented COVID19 negative testing prior to procedure.
  Interventions: Procedure: Major surgery involving general anesthesia

INTERVENTIONS:
Procedure: Major surgery involving general anesthesia — EHR documented SAR-CoV-2 PCR nasopharyngeal swab results confirming Covid-19 status within one year of undergoing surgical procedure at Kern Medical Center.
  Other Names: Diagnostic Test: SAR-CoV-2 PCR nasopharyngeal swab

SUMMARY:
Following the introduction of the COVID-19 vaccination, elective surgeries have resumed, allowing for greater insight into the postoperative period and outcomes aims on-going COVID-19 infections. This study aimed to evaluate risk factors of postoperative morbidity and mortality in patients who had surgery within one year of testing positive for COVID-19.

DETAILED DESCRIPTION:
SARS-CoV-2 (COVID-19) has infected over 100,000,000 million people in the United States (US). During the "first wave" in the US, medical facilities were advised to limit operative exposure, stratify operative cases by both risk and urgency and cancel elective procedures.

With over 60% of the US population considered fully vaccinated as of May of 2020, elective surgeries resumed amid periodic outbreaks allowing for continued insight into the impact of COVID-19 on the postoperative recovery process. However, relative to the volume of data on active infections, there is far less concerning the sequelae of previous infections. Therefore, the purpose of this study is to analyze a safety net hospital's experience regarding postoperative complications in patients that underwent surgical procedures requiring general anesthesia within a year of testing positive for COVID-19.

This is a retrospective study from a high-volume tertiary referral center and safety net hospital in Bakersfield, California. After approval by the Institutional Review Board, the electronic health record (EHR) was queried for all positive COVID-19 patients that underwent a surgical procedure of any kind requiring general anesthesia from 5 May 2020 to 31 December 2022. A total of 7,696 patients met inclusion criteria. 420 tested positive for COVID-19. Participants were subdivided into three study groups defined as symptomatic COVID-19 infection, asymptomatic COVID-19 infection, and COVID-19 negative control group.

Individual chart review allowed for subclassification based on symptomatology, admission status, length of admission, American Society of Anesthesiologist Physical Status Classification System (ASA), qSOFA and GCS rating along with COVID-19 and surgical complications Patients were required to have a COVID-19 diagnosis within one year of surgery. Categorical variables assessed in participants included age, sex, BMI, race, ICU or DOU stay. Post-operative complications assessed for included hospital length of stay, 30-day mortality, 30-day readmission, cardiac arrest, septic shock, acute kidney injury, acute respiratory distress syndrome, deep vein, thrombosis, pulmonary embolism, respiratory failure and pneumonia.

Statistical analysis was completed by the institution's statistician. Using Fisher extract, ANOVA, univariate and multivariate logistic regression analyses, odds ratios and p-values were obtained to evaluate for statistically significant correlations between categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Documented SAR-CoV-2 PCR nasopharyngeal swab within 1 year of major surgical intervention requiring general anesthesia

Exclusion Criteria:

* Surgical procedures using solely MAC and/or local anesthesia. Additionally, percutaneous endoscopic gastrostomy tube placements were omitted.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants who presented to Kern Medical Center, a high-volume tertiary referral center and safety net hospital located in Bakersfield, California between May 2020 to December 2022, who underwent a surgical procedure requiring general anesthesia. Participants were required to have a EHR documented SAR-CoV-2 PCR nasopharyngeal swab within one preoperatively.
  Study excludes surgical procedures using only MAC or local anesthesia as well as percutaneous endoscopic gastrostomy tube placement.
  A total of 7,696 patients were included, 420 tested positive for COVID-19 (7.6% were symptomatic and 4.8% were asymptomatic) and 7,276 tested negative (10.9% qualified as control).
Sampling Method: Non-Probability Sample
Enrollment: 7696 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Surgical complication rate | 05/05/2020-12/01/2022
  Post operative morbidity and mortality rate

CONTACTS AND LOCATIONS:
Locations (1):
- Kern Medical Center, Bakersfield, California, United States

IPD SHARING:
Plan to Share IPD: No